CLINICAL TRIAL: NCT06776757
Title: Sintilimab in Combination with Cetuximab and Chemotherapy As First-line Treatment for RAS/BRAF Wild-type Advanced Colorectal Cancer: an Open-label, Non-comparative, Phase 1b/2 Dose Escalation and Expansion Trial
Brief Title: Sintilimab in Combination with Cetuximab and Chemotherapy As First-line Treatment for RAS/BRAF Wild-type Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YW2023-25-2
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Sintilimab, Cetuximab, Chemotherapy, first-line, mCRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1b Dose Exploration (Experimental): Cetuximab and chemotherapy dose fixed, Sintilimab dose escalation to determine maximum tolerated dose in patients with RAS/BRAF wild-type mCRC
  Interventions: Drug: Sintilimab+Cetuximab+Chemotherapy (mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI)
- Phase 2 Expansion (Experimental): Phase 2 evaluation of the clinical activity of intilimab in combination with Cetuximab and chemotherapy in patients with RAS/BRAF wild-type mCRC
  Interventions: Drug: Sintilimab+Cetuximab+Chemotherapy (mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI)

INTERVENTIONS:
Drug: Sintilimab+Cetuximab+Chemotherapy (mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI) — Sintilimab (100mg,150mg, 200mg; Q3W) +Cetuximab (500mg/m²,Q2W)+Chemotherapy（mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI）
  Arms: Phase 1b Dose Exploration
Drug: Sintilimab+Cetuximab+Chemotherapy (mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI) — Sintilimab (Based on Phase 1b recommended dose; Q3W) +Cetuximab (500mg/m²,Q2W)+Chemotherapy（mFOLFOX6/FOLFIRI/CAPEOX/CAPIRI）
  Arms: Phase 2 Expansion

SUMMARY:
In 2018, global cancer incidence reached 18.1 million new cases, with 9.6 million cancer-related deaths. Colorectal cancer ranked as the third most common malignancy by incidence. Data from the U.S. NIH SEER database indicate a five-year survival rate for colorectal cancer of approximately 65%. Specifically, the survival rate is 90% for localized (non-metastatic) cases, 71% for regional (lymph node metastasis) cases, and only 14% for advanced metastatic cases. According to the China Society of Clinical Oncology (CSCO) guidelines, first-line therapy for advanced colorectal cancer typically involves chemotherapy combined with targeted agents, such as bevacizumab or cetuximab, yielding a median survival of 20-30 months. Prognosis is generally better for RAS wild-type patients compared to those with RAS mutations. In subsequent lines of therapy, chemotherapy combined with targeted therapy results in remission for approximately 22% of patients, although overall survival rarely exceeds 12 months.

Basic research has demonstrated that cetuximab, when combined with chemotherapy, enhances the infiltration of NK cells, cytotoxic T cells, and other immune cells into the tumor microenvironment. In head and neck cancer, an increase in PD-1+ and TIM-3+ tumor-infiltrating lymphocytes (TILs) during cetuximab treatment was negatively correlated with treatment response. Blocking these immune checkpoints may improve cetuximab-based immunotherapy by reversing CD8+ TIL dysfunction, potentially enhancing clinical outcomes. The cetuximab-chemotherapy regimen increases tumor immunogenicity by inducing tumor cell death and antigen release. When combined with immune checkpoint inhibitors, cetuximab may convert "cold tumors" into "hot tumors," thus synergistically improving tumor cell elimination. Additionally, cetuximab has been shown to activate tumor-promoting M2 macrophages, particularly CD163-positive macrophages in colorectal cancer, which produce high levels of Fc-γ receptors and PD-L1, supporting the theoretical basis for combining cetuximab with immune checkpoint inhibitors in colorectal cancer treatment.

In patients with locally advanced colorectal cancer, immune checkpoint inhibitors like PD-1 and CTLA-4 inhibitors have shown preliminary efficacy. The NICHE study reported a 100% pathological response in MSI-H patients and a 27% response in MSS-type patients, indicating potential benefits and safety of immunotherapy in both MSI-H sensitive and MSS/pMMR populations. For first-line treatment of advanced colorectal cancer, the BBCAPX Phase II study showed that sintilimab combined with CapeOX and bevacizumab resulted in an objective response rate (ORR) of 84% and a 100% disease control rate in RAS-mutant, MSS-type metastatic colorectal cancer (mCRC) patients. Similarly, the AIO-KRK-0216 study found that a combination of Avelumab (PD-L1), cetuximab, and chemotherapy produced an ORR of 79.5% in first-line MSS-type metastatic colorectal cancer. In later-line therapy, the REGONIVO Phase II study reported a 36% ORR for PD-1 monoclonal antibody combined with anti-angiogenesis agents (chemotherapy, targeted therapy) in metastatic colorectal cancer, with a 33% ORR for MSS-type patients. The median progression-free survival (PFS) was 7.9 months, though median overall survival (OS) had not been reached.

ELIGIBILITY:
Inclusion Criteria:

1.Sign a written informed consent before implementing any trial-related procedures.

2.Age between 18 and 75 years old.

3.No gender restrictions.

4.Histologically or cytologically confirmed inoperable or recurrent metastatic colorectal cancer (AJCC 8th edition, Stage IV).

5.No prior systemic antitumor treatment, or at least 6 months since the completion of adjuvant therapy.

6.At least one measurable lesion as per the RECIST 1.1 criteria for solid tumors.

7.Tumor tissue with both RAS and BRAF mutations being wild-type. 8.Tumor tissue with PD-L1 CPS ≥1, TPS ≥1%, or CD8+ TILs ≥2%. 9.ECOG performance status score of 0 or 1. 10.Expected survival time >3 months. 11.Sufficient organ function and bone marrow compensation function are required, and the subjects must meet the following laboratory criteria:

1. .Neutrophil Absolute Count (ANC) ≥ 1.5 x 10^9/L, provided that granulocyte colony-stimulating factor has not been used in the past 14 days.
2. .Platelet count ≥ 90 x 10^9/L, provided that no blood transfusion has been received in the past 14 days.
3. .Hemoglobin > 9 g/dL, provided that no blood transfusion or erythropoiesis-stimulating agents have been used in the past 14 days.
4. .Total bilirubin ≤ 1.5× Upper Limit of Normal (ULN); or total bilirubin > ULN but direct bilirubin ≤ ULN.
5. .Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5× ULN (patients with liver metastasis are allowed to have ALT or AST ≤ ULN).
6. .Serum creatinine ≤ 1.5× ULN, and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 ml/min.
7. .Normal coagulation function, defined as International Normalized Ratio (INR) or prothrombin time (PT) ≤ 1.5× ULN.
8. .Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with normal total T3 (or FT3) and FT4 levels may also be included.
9. .Normal myocardial enzyme levels (subjects with isolated laboratory abnormalities that the investigator determines to have no clinical significance may still be eligible for inclusion). (Optional) 12.For female subjects of reproductive potential, a urine or serum pregnancy test must be performed within 3 days prior to the first dose of study medication (Cycle 1, Day 1), and the result must be negative. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non-reproductive-aged females are defined as those who are at least 1 year postmenopausal or have undergone surgical sterilization or hysterectomy.

13.If there is a risk of pregnancy, all subjects (male and female) must use a contraceptive method with a failure rate of less than 1% throughout the treatment period and for 120 days after the last dose of study drug (or for 180 days after the last dose of chemotherapy).

Exclusion Criteria:

1. Previously received chemotherapy, cetuximab, or other anti-EGFR targeted therapies;
2. Previously received any of the following therapies: anti-PD-L1, anti-PD-L2 drugs, or drugs targeting other stimulatory or co-inhibitory T cell receptors (e.g., CTLA-4, OX-40, CD137) (adjustable);
3. Symptomatic or high-risk conditions such as obstruction, bleeding, perforation, pneumonia (including non-infectious pneumonia treated with corticosteroids or ongoing pneumonia treatment);
4. Diagnosed with other malignant diseases outside of colorectal cancer within 5 years prior to the first dose (excluding surgically cured basal cell carcinoma, squamous cell carcinoma of the skin, and/or surgically resected carcinoma in situ);
5. Currently participating in an interventional clinical trial or received other investigational drugs or devices within 4 weeks prior to the first dose;
6. Received traditional Chinese medicine with antitumor indications or immune-regulating drugs (including thymosin, interferons, interleukins, excluding local use for pleural effusion) as systemic therapy within 2 weeks prior to the first dose;
7. Experienced an active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments;
8. Receiving systemic corticosteroid therapy (excluding nasal, inhaled, or other forms of localized corticosteroids) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug. Note: Physiological doses of corticosteroids (≤10 mg/day of prednisone or equivalent) are allowed;
9. Received blood transfusion within 7 days prior to the first dose of treatment;
10. Clinically uncontrolled pleural or peritoneal effusion (patients who do not require drainage or have stable effusion for 3 days after stopping drainage may be enrolled);
11. Known history of allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
12. Known allergy to the study drug, sindilizumab, chemotherapy, targeted drug active ingredients, or excipients;
13. Presence of multiple factors affecting oral drug absorption (e.g., difficulty swallowing, post-gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc.);
14. Not fully recovered from toxicity and/or complications caused by any previous interventions before starting treatment (i.e., ≤ Grade 1 or back to baseline, excluding fatigue or alopecia);
15. Known history of HIV infection (i.e., HIV 1/2 antibody positive).
16. Untreated active hepatitis B (defined as HBsAg positive with detectable HBV-DNA copy numbers greater than the normal value upper limit in the testing laboratory of the research center); Note: Hepatitis B patients who meet the following criteria may also be included:

1).HBV viral load <1000 copies/ml (200 IU/ml) before the first dose; the participant should receive anti-HBV treatment throughout the study chemotherapy period to prevent viral reactivation.

2).For participants who are anti-HBc (+), HBsAg (-), anti-HBs (-), and have a negative HBV viral load, prophylactic anti-HBV treatment is not required, but close monitoring for viral reactivation is necessary.

17.Active HCV infection (HCV antibody positive and HCV-RNA level above the detection limit).

18.Vaccination with live vaccines within 30 days before the first dose (Cycle 1, Day 1); Note: An inactivated seasonal flu vaccine is allowed within 30 days prior to the first dose. However, intranasal live attenuated flu vaccines are not permitted.

19.Pregnant or breastfeeding women. 20.Presence of any serious or uncontrolled systemic diseases, such as:

1. .Significant and symptomatic abnormalities in rhythm, conduction, or morphology on resting electrocardiogram that are difficult to control, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation;
2. .Unstable angina, congestive heart failure, or chronic heart failure with New York Heart Association (NYHA) classification ≥ 2.
3. .History of any arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accidents, or transient ischemic attacks (TIA), etc.;
4. .Poorly controlled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
5. .History of non-infectious pneumonia requiring corticosteroid treatment within 1 year prior to the first dose, or currently has clinically active interstitial lung disease;
6. .Active pulmonary tuberculosis;
7. .Presence of active or uncontrolled infections requiring systemic treatment;
8. .Presence of clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction;
9. .Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. .Poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L);
11. .Urinalysis showing urine protein ≥ ++, and confirmed 24-hour urine protein quantification > 1.0 g;
12. .Presence of psychiatric disorders that prevent the patient from cooperating with the treatment; 21.A history or evidence of diseases that may interfere with the trial results, hinder the subject's full participation in the study, abnormal treatment or laboratory test values, or any other situation the investigator deems unsuitable for inclusion, including potential risks considered by the investigator that would make the participant unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 6 months
  The objective response rate is estimated by the proportion (percentage) of participants with the best response of complete response (CR), or partial response (PR) by RECIST 1.1 criteria, with corresponding exact 95% confidence limits being reported.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 12 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, National Clinical Research Center for Cancer, Cancer Hospital & Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided